CLINICAL TRIAL: NCT04277455
Title: Effect of Ultrasound Guided Laser Ablation Therapy on Symptomatic Benign Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson Thomas (Other)
Collaborators: Mercy Research (Other)
Responsible Party: Sponsor-Investigator, Johnson Thomas, Principal Investigator, Mercy Research
Organization: Mercy Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-113
Record Dates: First submitted 2020-02-11; First posted 2020-02-20 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Nodule
Keywords: Benign thyroid nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment arm (Experimental): Patients will receive laser treatment for benign symptomatic nodules
  Interventions: Device: Laser ablation of benign thyroid nodule

INTERVENTIONS:
Device: Laser ablation of benign thyroid nodule — Ablating symptomatic benign thyroid nodules using laser

SUMMARY:
This is a prospective trial to evaluate the effects of laser ablation on symptomatic benign thyroid nodules. The study is designed to assess the clinical efficacy, safety, tolerability and impact on symptoms of single ultrasound guided laser ablation treatment of symptomatic benign thyroid nodules. Approximately 20 subjects will undergo laser ablation of symptomatic benign nodules.

DETAILED DESCRIPTION:
* Laser ablation will be carried out in a single session under sterile conditions and ultrasound guidance with the support of Echolaser Smart Interface.
* Local anesthesia will be offered.
* The treatment plan will be assisted using the Echolaser Smart Interface.
* Depending on the shape and volume of the nodule to be treated, the investigator will determine whether one or two needles positioned parallel to each other along the longitudinal axis of the nodule will need to be used for treatment.
* Under ultrasound guidance, the investigator will introduce up to two 21-gauge introducer needles through the Guide kit into the target thyroid lesion percutaneously.
* Once the correct positioning of the needles has been verified under ultrasound imaging, an optical fiber is introduced into each needle with its tip protruding 5 mm out of the needle and in direct contact with the tissue to be ablated.
* Laser beam emission through the flat-tipped optical fiber produces a lesion (coagulation volume) within the nodule of an ellipsoidal shape, one third of which is positioned behind the tip of the fiber, and two-thirds in front.
* Each application session will last between 400 and 600 seconds under a laser source power output of 3W. An application is defined as the time between turning on and turning off the laser source.
* Up to 3 applications may be carried out during the same treatment session by pulling back along the needle and fiber axis by 0.5-1.0-1.5 cm to allow for treatment of tissue area not treated with previous application.
* Following completion of the laser ablation, the fibers will be removed followed by extraction of the needle(s). Hemostasis will be achieved at the site of needle insertion by applying pressure to the site.
* External bleeding will be assessed by visual inspection following extraction of the needle.
* Internal bleeding and potential nodule rupture will be assessed by ultrasound of the thyroid/neck with doppler flow assessment by the investigator following needle extraction using GE Logiq P6 ultrasound.The site will be covered with a sterile dressing/bandage.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, Age ≥18 years
* Thyroid Stimulating Hormone (TSH) within normal limits
* Presence of thyroid nodule >29 mm and ≤60 mm in the longest dimension on ultrasound imaging
* Symptoms from thyroid nodule - tightness or pressure in neck, neck tenderness, neck pain, difficulty swallowing, voice changes, shortness of breath or cosmetic disfigurement
* Solid thyroid nodule with less than 20% cystic component
* Cytological benign nodule proven by previous biopsy within 2 years
* Ability to place the laser tip inside the nodule and to keep vital structures (i.e. trachea and esophagus) outside the zone of injury. To achieve this safe zone, we will leave a minimum of 17 mm distance between the fiber tip anterior to the vital structures and 10 mm from the fiber tip in all other dimensions.
* Not on anticoagulants or anticoagulants stopped for appropriate amount of time based on the pharmacology of the drug
* Ability to understand and willingness to provide informed consent

Exclusion Criteria:

* Pregnancy
* Diagnosis of Hyperthyroidism
* Malignant thyroid nodule
* Egg shell or coarse calcification in the thyroid nodule
* Patient on anticoagulation which cannot be stopped due to medical reasons
* Coagulopathy
* Thyroid nodules in contact with trachea, esophagus or major blood vessels
* Prior neck surgery
* Prior radiation to head and neck
* Previous radioactive iodine treatment
* Current iodine supplementation
* Current anti-thyroid medication
* Biotin supplementation within 2 days prior to enrollment
* Allergy to Ethyl chloride spray or lidocaine
* Physical and psychological conditions that prevent safe administration of the procedure as determined by the investigator
* Adults not able to consent
* Prisoners
* Individuals who cannot read and understand English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Thomas, MD, FACE, Principal Investigator — Mercy Research
Locations (1):
- Mercy Clinic Endocrinology - Smith Glynn Callaway, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- [Background] Pacella CM, Mauri G, Achille G, Barbaro D, Bizzarri G, De Feo P, Di Stasio E, Esposito R, Gambelunghe G, Misischi I, Raggiunti B, Rago T, Patelli GL, D'Este S, Vitti P, Papini E. Outcomes and Risk Factors for Complications of Laser Ablation for Thyroid Nodules: A Multicenter Study on 1531 Patients. J Clin Endocrinol Metab. 2015 Oct;100(10):3903-10. doi: 10.1210/jc.2015-1964. Epub 2015 Aug 14. PMID 26274342
- [Background] Papini E, Rago T, Gambelunghe G, Valcavi R, Bizzarri G, Vitti P, De Feo P, Riganti F, Misischi I, Di Stasio E, Pacella CM. Long-term efficacy of ultrasound-guided laser ablation for benign solid thyroid nodules. Results of a three-year multicenter prospective randomized trial. J Clin Endocrinol Metab. 2014 Oct;99(10):3653-9. doi: 10.1210/jc.2014-1826. Epub 2014 Jul 22. PMID 25050903
- [Background] Pacella CM, Mauri G, Cesareo R, Paqualini V, Cianni R, De Feo P, Gambelunghe G, Raggiunti B, Tina D, Deandrea M, Limone PP, Mormile A, Giusti M, Oddo S, Achille G, Di Stasio E, Misischi I, Papini E. A comparison of laser with radiofrequency ablation for the treatment of benign thyroid nodules: a propensity score matching analysis. Int J Hyperthermia. 2017 Dec;33(8):911-919. doi: 10.1080/02656736.2017.1332395. Epub 2017 Jun 12. PMID 28605944

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 56 [34 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline volume of the index thyroid nodule [Mean (Full Range); unit: mm^3] | 17.43 [5.51 to 28.22]
Baseline visual inspection of the neck at 1 m [Number; unit: participants]
  Presented with visible nodule at a distance of > 1 meter | 10
  Presented with no visible nodule at a distance of > 1 meter | 0
Baseline symptoms [Number; unit: participants]
  Reported neck pain | 1
  Reported neck tenderness | 6
  Reported neck tightness | 9
  Reported difficulty swallowing | 7
  Reported voice changes | 2
  Reported shortness of breath | 2
  Reported cosmetic disfigurement | 5
Baseline TSH [Mean (Full Range); unit: µU/mL] | 1.22 [0.29 to 2.01]
Baseline Free T4 [Mean (Full Range); unit: ng/dL] | 1.26 [1.02 to 1.56]
Baseline Free T3 [Mean (Full Range); unit: pmol/L] | 3.12 [2.60 to 3.90]
Baseline antithyroid antibodies [Median (Full Range); unit: IU/mL]
  TPO Antibodies | 6.8 [1.000 to 29.000]
  Thyroglobulin Antibodies | 11 [.0001 to 921]
Baseline status of vocal fold structure and function [Count of Participants; unit: Participants]
  Presented as normal | 10
  Presented as abnormal | 0
Baseline pain score [Number; unit: participants] — Pain score rating from 1-10 was used with "1" being minimal discomfort and "10" indicating the worst possible pain.
  participants
    Pain score of 0 | 6
    Pain score of 1 | 2
    Pain score of 4 | 2
Cosmetic assessment at baseline [Mean (Full Range); unit: score on a scale] — Patients perceived cosmetic appearance will be measured using a numerical scale at baseline, immediately after procedure and then at 3,6 and 12 months after procedure using following question. On a scale from 0 to 10, how much does your thyroid nodule affect your appearance? 0 being the best outcome and 10 being the worst outcome.
  score on a scale | 2.7 [0 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Change in Radiographic Volume of Thyroid Nodule From Baseline at 3, 6 and 12 Months After Laser Ablation
Description: Percentage change from baseline volume will be calculated at 3, 6 and 12 months after laser treatment.
Time Frame: 12 months
Population: 9 subjects completed the 12-month post-procedure study visit. One patient did not return for the 12-month follow up visit and was determined to be lost to follow-up.
Measure: Mean (Full Range); unit: percentage of volume reduction
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
percentage of volume reduction
  Average change in volume of thyroid nodule at the 3-months post-procedure study visit | 63.4 [26.3 to 75.5]
  Average change in volume of thyroid nodule from baseline to 12-months: number analyzed (Participants) | 9
  Average change in volume of thyroid nodule from baseline to 12-months | 71.087 [30.95 to 91.062]

2. Primary Outcome: Change in the Thyroid Function After Laser Treatment Assessed by the Measurement of TSH and Free T4 at 3, 6 and 12 Months After Laser Ablation
Description: Number of patients who develops hypo or hyperthyroidism 3,6 and 12 months after laser treatment.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
participants
  Demonstrated a clinically significant change | 0
  Did not demonstrate a clinically significant change | 10

3. Primary Outcome: Change in Doppler Grade at 3, 6, and 12 Months After Laser Ablation
Description: Number of patients who had changes in blood flow inside the thyroid nodule as evidenced by change in Doppler grade.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Participants
  3 months | 1
  6 months | 0
  12 months: number analyzed (Participants) | 9
  12 months | 0

4. Primary Outcome: Change in Thyroid Antibody Levels 3,6 and 12 Months After Laser Ablation
Description: Number of patients who develops new thyroid antibodies 3,6, and 12 months after laser ablation
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
participants
  Demonstrated a clinically significant change | 0
  Did not demonstrate a clinically significant change | 10

5. Primary Outcome: Cosmetic Assessment at 3,6 and 12 Months and Immediately After Laser Ablation Measured Using a Numerical Scale
Description: Patients perceived cosmetic appearance will be measured using a numerical scale at baseline, immediately after procedure and then at 3, 6 and 12 months after procedure using following question. On a scale from 0 to 10, how much does your thyroid nodule affect your appearance? 0 being the best outcome and 10 being the worst outcome.
Time Frame: 3 months, 6 months, and 12 months after procedure
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
score on a scale
  Reported Immediately after procedure | 3 [0 to 7]
  3 months | 0.9 [0 to 3]
  6 months | 0.6 [0 to 3]
  12 months: number analyzed (Participants) | 9
  12 months | .78 [0 to 3]

6. Secondary Outcome: Reported Pain Score on the Numerical Scale Immediately Post Procedure.
Description: Change in pain will be measured using a numerical scale at baseline, immediately post procedure and 3 months after procedure using the following question. Rate your pain on a scale from 0 to 10 where 0 is no pain and 10 is the worst pain possible.
Time Frame: Immediately post-procedure
Measure: Mean (Full Range); unit: pain score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 9
pain score on a scale | 5.5 [2 to 9]

7. Secondary Outcome: Tolerability of Ultrasound Guided Percutaneous Laser Ablation for Treatment of Symptomatic Benign Thyroid Nodules as Reported Through a Questionnaire After the Procedure.
Description: Participants will be asked to answer the following questionnaire after the procedure.
  How likely is it that you would have the laser ablation procedure again? 1 = Very Likely 2 = Somewhat Likely 3 = Not Likely
Time Frame: Post-procedure on the day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Participants
  1 = Very Likely | 7
  2 = Somewhat Likely | 3
  3 = Not Likely | 0

8. Secondary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed by CTCAE v4.0
Description: Treatment related adverse events will be captured using CTCAE v4,0 format
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Participants
  Feeling of a knot in neck at needle stick site | 1
  Sensation of lump in throat | 1
  Burning sensation in neck at needle stick site | 1
  Sore throat | 1
  Coughing | 1
  Bruising to neck | 2
  Pain/discomfort with swallowing | 2
  Difficulty swallowing | 1
  Swelling at needle stick site | 6
  Pain/soreness in neck | 10

9. Secondary Outcome: Reported Pain Score on the Numerical Scale 3 Months Post Procedure.
Description: as for outcome 6
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
participants
  Pain score of 0 | 10
  Pain score greater than 0 | 0

10. Secondary Outcome: Tolerability of Ultrasound Guided Percutaneous Laser Ablation for Treatment of Symptomatic Benign Thyroid Nodules as Reported Through a Questionnaire After the Procedure.
Description: Participants will be asked to answer the following questionnaire after the procedure.
  How satisfied were you with the length of the laser ablation procedure? 1= Satisfied 2 = Neither 3 = Dissatisfied
Time Frame: Post-procedure on day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Participants
  1= Satisfied | 7
  2 = Neither | 2
  3 = Dissatisfied | 1

11. Secondary Outcome: Tolerability of Ultrasound Guided Percutaneous Laser Ablation for Treatment of Symptomatic Benign Thyroid Nodules as Reported Through a Questionnaire After the Procedure.
Description: Participants will be asked to answer the following questionnaire after the procedure.
  How much discomfort did you have with the laser ablation procedure? 1= Less than I thought 2 = About what I thought 3 = More than I thought
Time Frame: Post-procedure on day of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 10
Participants
  1= Less than I thought | 1
  2 = About what I thought | 3
  3 = More than I thought | 6

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study, an average of 12 months.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=10)
Feeling of a knot in neck at needle stick site (Skin and subcutaneous tissue disorders) | 1
Sensation of lump in throat (Musculoskeletal and connective tissue disorders) | 1
Burning sensation in neck at needle stick site (Skin and subcutaneous tissue disorders) | 1
Sore throat (Musculoskeletal and connective tissue disorders) | 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 1
Bruising to neck (Skin and subcutaneous tissue disorders) | 2
Pain/discomfort with swallowing (Musculoskeletal and connective tissue disorders) | 2
Difficulty swallowing (Musculoskeletal and connective tissue disorders) | 1
Swelling at needle stick site (Skin and subcutaneous tissue disorders) | 6
Pain/soreness in neck (Musculoskeletal and connective tissue disorders) | 10

LIMITATIONS AND CAVEATS:
There are a few limitations to this study. This is a single-center study with a small sample size, which makes findings less generalizable. Pain, tolerability, and cosmetic assessments are subjective and hard to quantify objectively. Hence, we used standardized scales to reduce subjectivity. There was also no control group. Longterm outcomes were not assessed because subjects were only followed for 12 months after the laser ablation procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04277455/Prot_SAP_001.pdf